CLINICAL TRIAL: NCT07345936
Title: Endoscopic Treatment of Post Surgical Biliary Tract Injury
Acronym: EpSB
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9943
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Biliary Tract Injuries
Keywords: Biliary tract injuries; Endoscopic treatment; Iatrogenic injuries of the bile ducts

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to determine the technical and clinical success rate of endoscopic treatment in a population presenting only with iatrogenic injuries of the bile ducts, excluding the cystic duct.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old)
* Subject who has had a wound of the common bile duct or intrahepatic bile ducts following hepatobiliary surgery (laparotomy or laparoscopic cholecystectomy or major or minor hepatectomy)
* Subject treated in one of the associated centers between January 1, 2021, and December 31, 2024

Exclusion Criteria:

* Biliary wound occurring on a long cystic duct or gallbladder stump during partial cholecystectomy.
* Biliary leakage complicating liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient who has had a wound of the common bile duct or intrahepatic bile ducts following hepatobiliary surgery (laparotomy or laparoscopic cholecystectomy or major or minor hepatectomy)
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04-17 (Estimated)

PRIMARY OUTCOMES:
Clinical success rate of the initial endoscopic procedure | Immediately after surgery
  Success rate:
  This is the percentage of patients for whom the treatment was successful Expressed as a percentage.
  Example:
  Out of 100 patients, if 85 improve, the success rate is 85%.
Clinical success rate at 3 months after the end of treatment | 3 months after the end of treatment
  Success rate:
  This is the percentage of patients for whom the treatment was successful Expressed as a percentage.
  Example:
  If 100 patients are treated and 80 improve, the success rate is 80%.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Hépato-gastroentérologie - CHU de Strasbourg - France, Strasbourg, France